CLINICAL TRIAL: NCT03417531
Title: Sarcopenia Prevention With a Targeted Exercise and Protein Supplementation Program
Acronym: STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); University Hospital, Zürich (Other); University Geriatric Medicine Felix Platter, Basel, Switzerland (Unknown); Omanda AG, Baar, Switzerland (Unknown); Ferrari Data Solution (Other); City Hospital Waid and Triemli, Zurich, Switzerland (Unknown); Cantonal Hospital of St. Gallen (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-02045
Record Dates: First submitted 2018-01-09; First posted 2018-01-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Frailty; Malnutrition; Protein; Fall
Keywords: Protein supplementation; Home exercise program; Falls prevention; Seniors; Autonomy
MeSH Terms: conditions — Sarcopenia; Frailty; Kwashiorkor | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Protein Supplement plus Active Exercise (Active Comparator): Participants will ingest twice daily 23.7 g of L-leucine-enriched whey protein isolate powder (equivalent to 20 g of Protein) and perform a simple home exercise strength program (3x30 minutes/week)
  Interventions: Dietary Supplement: Protein Supplement; Procedure: Active Exercise
- Protein-free Supplement plus Active Exercise (Active Comparator): Participants will ingest twice daily 23.7 g of a protein-free, isocaloric powder blend and perform a simple home exercise strength program (3x30 minutes/week)
  Interventions: Dietary Supplement: Protein-free Supplement; Procedure: Active Exercise
- Protein Supplement plus Control Exercise (Active Comparator): Participants will ingest twice daily 23.7 g of L-leucine-enriched whey protein isolate powder (equivalent to 20 g of Protein) and perform a joint flexibility home exercise program (3x30 minutes/week)
  Interventions: Dietary Supplement: Protein Supplement; Procedure: Control Exercise
- Protein-free Supplement plus Control Exercise (Sham Comparator): Participants will ingest twice daily 23.7 g of a protein-free, isocaloric powder blend and perform a joint flexibility home exercise program (3x30 minutes/week)
  Interventions: Dietary Supplement: Protein-free Supplement; Procedure: Control Exercise

INTERVENTIONS:
Dietary Supplement: Protein Supplement — Predosed protein powder; can be added to various dishes and drinks
  Other Names: Moltein® Ready-to-Shake
  Arms: Protein Supplement plus Active Exercise; Protein Supplement plus Control Exercise
Dietary Supplement: Protein-free Supplement — Predosed protein-free powder; can be added to various dishes and drinks
  Arms: Protein-free Supplement plus Active Exercise; Protein-free Supplement plus Control Exercise
Procedure: Active Exercise — Program includes five strength exercises that can be easily performed at home
  Arms: Protein Supplement plus Active Exercise; Protein-free Supplement plus Active Exercise
Procedure: Control Exercise — Program includes five flexibility exercises that can be easily performed at home
  Arms: Protein Supplement plus Control Exercise; Protein-free Supplement plus Control Exercise

SUMMARY:
Physical inactivity and protein malnutrition have been implicated to be key and modifiable causes of enhanced muscle mass loss among seniors. However, the individual benefit, as well as the additive or possibly interactive benefit of exercise and Protein supplementation on fall prevention has yet to be confirmed in a large clinical trial. This study aims to test the individual and combined effect and cost-effectiveness of a simple home exercise program and / or protein supplementation on the risk of falling in seniors at high risk of progressive muscle mass loss and sarcopenia.

DETAILED DESCRIPTION:
The number of seniors age 75 and older is predicted to double by 2030, as is the number of seniors with mobility disability, physical frailty and resulting consequences, such as falls and loss of autonomy. This causes an enormous challenge to the individual, to medical care, and the society as a whole. A condition that is considered central to the development of physical frailty and its consequences is sarcopenia, the loss of muscle mass and strength. To date sarcopenia is underdiagnosed in clinical care and effective treatments for sarcopenia are missing.

This study aims to test the individual and combined effect and cost-effectiveness of a simple home exercise program and / or protein supplementation on the risk of falling in seniors at high risk of progressive muscle mass loss and sarcopenia.

The STRONG trial will be a 2x2 factorial design multi-centre double-blind randomized controlled clinical trial among 800 senior men and women; study duration is 12 months. The primary endpoint is the rate of falling. Key secondary endpoints include functional decline, and the proportion of seniors with frailty, sarcopenia, and loss of autonomy. STRONG will further assess the cost-effectiveness of the interventions based on health care utilization data collected every 2 months from each participant and observed incidence of the endpoints. Mechanistic endpoints include change in muscle mass by DXA(arms and legs), change in myostatin levels, and muscle quality (based on MRI).

The interventions are (1) a simple home exercise program (a validated strength-enhancing or a control joint flexibility exercise program) to be performed 3x30 minutes/week; and (2) protein supplementation (either 20g of whey protein or isocaloric powder given in two portions for breakfast and dinner each day). All participants will receive a control dose of 24'000 IU vitamin D per month (equivalent to 800 IU vitamin D/day) to ensure that over 97% of STRONG participants will be vitamin D replete (25-hydroxyvitamin D > 20 ng/ml) during the course of the trial.

The trial will have clinical visits at baseline, 6 months, and 12 months. In between clinical visits, telephone interviews will be performed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 of 5 frailty criteria, definition by Linda Fried: 1) weight loss of > 4.5 kg in the last 12 months; 2) reduced grip strength in Martin Vigorimeter test: ♂ ≤ 64 kPa, ♀ ≤ 42 kPa; 3) standardized question on exhaustion as published by Fried et al.; 4) gait speed < 1 m/s; 5) 6-minute walk test < 300 meters and/or Injurious (any injury) low trauma fall in the last 12 months prior to enrollment
* Reduced protein intake defined as a score ≤ 0.5 at item K of the Mini Nutritional Assessment (MNA)
* Community-dwelling or assisted living

Exclusion Criteria:

* Mini-mental state examination (MMSE) < 24 (inability to follow the study procedures and give written informed consent)
* Inability to come to the trial centers
* Inability to walk at least 3 meters with or without walking aid
* Severe kidney impairment (Glomerular filtration rate [GFR] < 30 ml/min)
* Inability to follow exercise instruction or inability to take protein powder mixed in drink or food (test at baseline screening examination)
* Severe gait impairment or diseases with a risk of recurrent falling (due to conditions such as, e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope)
* Major visual or hearing impairment or other serious illness that would preclude participation (e.g. alcohol abuse, alcoholic disease)
* Inability to read/speak/write in German (necessary to follow instructions incl. STRONG exercise manual)
* Living in a nursing home
* Contraindication to treatment (e.g. allergy)
* Contraindication to the vitamin D standard of care therapy

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 801 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Rate of falling | 12 months
  The circumstances and injuries associated with the fall will be ascertained with a questionnaire.

SECONDARY OUTCOMES:
Functional decline (change in lower extremity function) | Baseline, 6, and 12 months
  will be assessed with the Short Physical Performance Battery (SPPB)
Proportion of seniors with any falls and injurious falls | every 2 months over 12 months
  using the same method as for the primary endpoint
Proportion of seniors with established frailty | Baseline, 6, and 12 months
  Frailty will be defined as 3 out of the following 5 criteria are met: 1) weight loss of > 4.5 kg in the last 12 months; 2) reduced grip strength in Martin Vigorimeter test: ♂ ≤ 64 kPa, ♀ ≤ 42 kPa; 3) standardized question on exhaustion as published by Fried et al.; 4) gait speed < 1 m/s; 5) 6-minute walk test < 300 meters
Proportion of seniors with sarcopenia | Baseline, 6, and 12 months
  will be assessed both with the Baumgartner definition (muscle mass alone) and the European Working Group definition by Cruz-Jentoft24 (composite definition of muscle mass and impaired grip strength or gait speed)
Proportion of seniors admitted to nursing homes (loss of autonomy) | every 2 months over 12 months
  participants will be asked at visits/phone calls
Change in gait speed | Baseline, 6, and 12 months
  Gait speed will be measured over a distance of 4 meters. The participants will be asked to walk in their usual pace
Change in reaction time | Baseline, 6, and 12 months
  Reaction time will be assessed with repeated chair stands (5 repeats as part of the SPPB)
Change in grip strength | Baseline, 6, and 12 months
  Measured with Martin Vigorimeter
Change in aerobic capacity | Baseline, 6, and 12 months
  Aerobic capacity will be assessed with the 6 minute walk test. A walked distance of < 300 m will be used as a frailty criteria
Change in muscle mass (arms and legs) | Baseline, 6, and 12 months
  will be measured with IDXA machines (intelligent dual x-ray absorptiometry by GE Healthcare)
Change in bone mineral density (hip and lumbar spine) | Baseline and 12 months
  will be measured with IDXA machines (intelligent dual x-ray absorptiometry by GE Healthcare)
Change in physical activity | Baseline, 6, and 12 months
  will be assessed by an excerpt from the Nurses' Health Study (NHS) questionnaire
Change in quality of life | Baseline, 6, and 12 months
  will be assessed using the German Version of EuroQuol EQ5D-3L questionnaire according to the Austrian reference scale

OTHER OUTCOMES:
Health care utilization | every 2 months over 12 months
  assessed with a simple questionnaire to collect health care utilization information prospectively (MD visit, PT visit, hospitalizations in acute care etc)
Myostatin | Baseline, 6, and 12 months
  Blood Sample Assessment: Myostatin
IGF-1 | Baseline, 6, and 12 months
  Blood Sample Assessment: Insulin-like growth factor-1
CRP | Baseline, 6, and 12 months
  Blood Sample Assessment: C-Reactive Protein
Kidney function | Baseline, 6, and 12 months
  Blood Sample Assessment: creatinine
25-hydroxyvitamin D | Baseline, 6, and 12 months
  Blood Sample Assessment: 25-hydroxyvitamin D
Fasting insulin levels | Baseline, 6, and 12 months
  Blood Sample Assessment: fasting insulin levels
Fasting blood glucose | Baseline, 6, and 12 months
  Blood Sample Assessment: fasting blood glucose
Change muscle quality (sub-sample of 140 participants) | Baseline and 12 months
  Assessed with whole Body MRI's in a subsample of f140 participants
Any non-vertebral fracture | every 2 months over 12 months
  All fractures will be confirmed by x-ray or medical record.
Mortality | every 2 months over 12 months
  will be assessed by personal contact
Rate of SAEs in general | over 12 months
  Serious Adverse Events
Rate of SAEs related to study intervention | over 12 months
  Serious Adverse Events
Adherence to intervention (dietary supplement) | Baseline, 6, and 12 months
  nitrogen excretion from 24-h/spot urine
Adherence to intervention (dietary supplement) | over 12 months
  will be assessed by questionnaire and diary
Adherence to intervention (exercise) | over 12 months
  will be assessed by questionnaire and diary
Covariate: Hearing | over 12 months
  will be assessed by a hearing test

CONTACTS AND LOCATIONS:
Overall Officials: Heike A. Bischoff-Ferrari, MD, DrPH, Principal Investigator — University of Basel
Locations (2):
- Switzerland (2):
  - University Geriatric Medicine Felix Platter, Basel, Basel, Basel
  - Centre on Aging and Mobility, University of Zurich and City Hospital Waid and Triemli, Zurich, Canton of Zurich